CLINICAL TRIAL: NCT02707939
Title: Observational Prospective Study on Behavioral Outcomes of Children With Autism Spectrum Disorder (ASD) in Comparison to Those Without Neurodevelopmental Diagnoses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Bistra Vlassakova, MD, Boston Children's Hospital
Other Study IDs: P00021473
Record Dates: First submitted 2016-03-10; First posted 2016-03-14 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Autism Spectrum Disorder; Anesthesia
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder: Patients with a diagnosis of autism spectrum disorder
  Interventions: Other: Observation
- Controls: Patients with no developmental diagnoses
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Patients will be observed before and after they receive anesthesia

SUMMARY:
Autism Spectrum Disorder (ASD) is the fastest growing neurodevelopmental disorder in the world. Approximately 1% of the population worldwide is affected by this disorder. Children with ASD exhibit some very stereo-typical behaviors. Their daily functionality depends on very rigid and predictable schedules and routines. Any changes in their schedules can often trigger negative emotional outbursts. The need to come to the hospital for procedures can be one such trigger. The purpose of this study is to examine the post anesthesia behavior outcomes of children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 2 years through 17 years of age scheduled for a procedure with anesthesia at Boston Children's Hospital
* Patients must have a diagnosis of Autism Spectrum Disorder (ASD) according to the DSM IV and DSM V (autism group) or an ASA score of I or II and no history of neurodevelopmental concerns (control group)

Exclusion Criteria:

-Families who are not able to read and speak English well enough to complete the validated surveys

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants with an ASD diagnosis and control patients who do not have any history of neurodevelopmental concerns who are scheduled for a procedure under anesthesia at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative behavioral changes in the participants | up to two weeks following anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Bistra Vlassakova, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arnold B, Elliott A, Laohamroonvorapongse D, Hanna J, Norvell D, Koh J. Autistic children and anesthesia: is their perioperative experience different? Paediatr Anaesth. 2015 Nov;25(11):1103-10. doi: 10.1111/pan.12739. Epub 2015 Sep 4. PMID 26338278
- [Background] Taghizadeh N, Davidson A, Williams K, Story D. Autism spectrum disorder (ASD) and its perioperative management. Paediatr Anaesth. 2015 Nov;25(11):1076-84. doi: 10.1111/pan.12732. Epub 2015 Aug 6. PMID 26248302
- [Background] van der Walt JH, Moran C. An audit of perioperative management of autistic children. Paediatr Anaesth. 2001 Jul;11(4):401-8. doi: 10.1046/j.1460-9592.2001.00688.x. PMID 11442855